CLINICAL TRIAL: NCT04216706
Title: Early Vascular Adjustments to Prevent Preeclampsia and Related Complications
Brief Title: Early Vascular Adjustments to Prevent Preeclampsia
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-4-118
Record Dates: First submitted 2019-12-19; First posted 2020-01-03 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2019-12

CONDITIONS: Preeclampsia; Small for Gestational Age at Delivery; HELLP Syndrome
Keywords: cardiac output; total peripheral vascular resistance; hemodynamic parameters; adaptation to pregnancy; tailored treatment
MeSH Terms: conditions — Pre-Eclampsia; HELLP Syndrome | interventions — Calcium Channel Blockers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tailored treatment advise in suboptimal adaptation: High-risk women admitted to a non-pregnant cardiovascular and cardiometabolic risk factor assessment are invited to participate in a follow-up program at four time-points during a subsequent pregnancy (i.e. at 12, 16, 20 and 30 weeks of gestational age). This program is additive to regular pregnancy check-ups, and all women are otherwise managed by their referring physicians. The aim of this program is to evaluate adaptation of maternal hemodynamic parameters in response to pregnancy, and to adjust deviant adaptation with tailored antihypertensive medication. Participation in this program is on voluntary basis, and not restricted to severity of complications in the first pregnancy.
  Interventions: Drug: tailored pharmaceutical treatment
- Care as usual during pregnancy: High-risk women admitted to a non-pregnant cardiovascular and cardiometabolic risk factor assessment who do not participate in the additional follow-up program.

INTERVENTIONS:
Drug: tailored pharmaceutical treatment — Tailored medication is advised in women with inadequate hemodynamic adaptation to pregnancy. Type of medication depends on total peripheral vascular resistance and heart rate. In short, women with a low peripheral vascular resistance in parallel with a high heart rate are advised a betablocker (labetalol), while a vasodilating agent (calcium channel blocker, nifedipine) was advised in women with a high total peripheral vascular resistance in combination with a low heart rate. Women with suboptimal adaptation to pregnancy without an extreme pronounced vascular profile are advised a centrally acting sympatholytic agent (methyldopa).
  Other Names: Betablocker; Centrally acting sympatholytic agent; Calcium channel blocker
  Groups: Tailored treatment advise in suboptimal adaptation

SUMMARY:
Women destined to develop gestational hypertensive complications often exhibit deviant hemodynamic adaptation patterns before overt clinical disease. Gestational hypertension and late onset preeclampsia are associated with an exaggerated rise in cardiac output on top of a higher prepregnant value, whereas a shallow rise in cardiac output and the lack of a peripheral resistance drop predisposes to the much less common early onset-preeclampsia along with impaired fetal growth. Early treatment of altered cardiac output and peripheral resistance adjustments might prevent development of gestational hypertensive complications. The investigators aim to evaluate early cardiovascular adjustments during pregnancy in a high-risk population, and to pharmaceutically adjust deviant cardiovascular adaptations with beta-blockade, centrally acting sympatholytic agents or vasodilating agents when appropriate to prevent adverse effects on neonatal birth weight.

DETAILED DESCRIPTION:
Healthy pregnancy is accompanied by major hemodynamic changes that benefit the uteroplacental circulation. A first-trimester drop in vascular resistance triggers several compensatory mechanisms, amongst an increase in blood volume and cardiac output, to maintain blood pressure. These adaptations continue and stand until delivery.

Women destined to develop gestational hypertensive complications often exhibit deviant hemodynamic adaptation patterns before overt clinical disease. On the one hand, gestational hypertension and late onset preeclampsia are associated with an exaggerated rise in cardiac output on top of a higher prepregnant value, whereas a shallow rise in cardiac output and the lack of a peripheral resistance drop predisposes to the much less common early onset-preeclampsia along with impaired fetal growth.

Antihypertensive therapy based on correction of the hemodynamic imbalance between cardiac output and peripheral resistance seems an effective strategy to improve blood pressure control in hypertensive pregnant women. Even more sophisticated, early treatment of altered cardiac output and peripheral resistance adjustments might prevent development of gestational hypertensive complications. One randomized controlled trial treated pregnant women with an augmented cardiac output with a selective beta-blocker, which resulted in a decreased prevalence of preeclampsia from 18% in the placebo group to 4% in the atenolol group (p = 0.04), at a cost of 440gram birth weight.

In line of this reasoning, the investigators aimed to evaluate early cardiovascular adjustments during pregnancy in a high-risk population (i.e. women with preeclampsia in their first pregnancy). In this health care traject, women with deviant adaptation to pregnancy were advised tailored medication, i.e. beta-blockade in women with an pronounced high cardiac output profile effectuated by a high heart rate, and a vasodilating agent in women with a high-resistance hemodynamic profile. Women with a mixed hemodynamic profile were advised a centrally acting sympatholytic agent. The investigators aimed to retrospectively compare outcome of women attending this health care project with women who received care as usual in their second pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* first pregnancy complicated by preeclampsia
* admitted to an extensive non-pregnant cardiovascular and metabolic risk factor assessment

Exclusion Criteria:

* women without an ongoing pregnancy after 24 weeks' gestational age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who had preeclampsia in their first pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Number of women that develop preeclampsia | during pregnancy, or up to 6 weeks after delivery
  Preeclampsia is defined as new-onset hypertension along with de novo proteinuria or other maternal organ dysfunction (i.e. renal insufficiency, liver involvement, neurological complications or hematological complications) after 20 weeks of gestation in previously normotensive women, or superimposed on chronic hypertension.

SECONDARY OUTCOMES:
Number of women that develop HELLP syndrome | during pregnancy, or up to 6 weeks after delivery
  HELLP-syndrome is defined as hemolysis (LDH > 600 U/L), elevated liver enzymes (AST -aspartate aminotransferase- and ALT -alanine aminotransferase- > 70 U/L) and low platelets (platelet count < 100.109/L)
Number of women that develop eclampsia | during pregnancy, or up to 6 weeks after delivery
  Seizures in women with preeclampsia
Number of women that have placental abruption during pregnancy | During pregnancy or at delivery
Stillbirth | during pregnancy until delivery
  Number of stillbirths in included women
Neonatal mortality | after delivery up to hospital discharge, which is assessed 6 weeks after due date of the mother
  Number of neonatal demise related to prematurity or as a consequence of maternal disease related to preeclampsia
Neonatal birth weight | measured at delivery
  birth weight of neonates
Neonatal birth weight centile | birth weight and other parameters measured at delivery
  Neonatal birth weight centile (adjusted for sex of neonate, gestational age at delivery and maternal parity)
Pregnancy outcome of women included | at delivery
  Gestational age at delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mulder EG, Ghossein-Doha C, Cauffman E, Lopes van Balen VA, Schiffer VMMM, Alers RJ, Oben J, Smits L, van Kuijk SMJ, Spaanderman MEA. Preventing Recurrent Preeclampsia by Tailored Treatment of Nonphysiologic Hemodynamic Adjustments to Pregnancy. Hypertension. 2021 Jun;77(6):2045-2053. doi: 10.1161/HYPERTENSIONAHA.120.16502. Epub 2021 Apr 5. PMID 33813842